CLINICAL TRIAL: NCT01230840
Title: Effect of Wheat Dextrin on Calcium and Magnesium Absorption
Acronym: Benefiber
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Laura Armas MD, Creighton University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 09-15249
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Colonic Inertia
Keywords: fiber; calcium; magnesium
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Control cookies will contain no wheat dextrin and will be taken 3 times daily for 2 weeks.
  Interventions: Dietary Supplement: placebo
- wheat dextrin (Experimental): wheat dextrin (formulated according to the supporter's established method), will be baked in cookies providing three doses per day (≈5 gram of wheat dextrin in each dose)for 2 weeks.
  Interventions: Dietary Supplement: wheat dextrin

INTERVENTIONS:
Dietary Supplement: wheat dextrin — 5 grams of wheat dextrin baked in cookies will be taken 3 times a day for 2 weeks
  Arms: wheat dextrin
Dietary Supplement: placebo — cookies not containing wheat dextrin will be taken 3 times a day for 2 weeks
  Arms: placebo

SUMMARY:
To compare calcium and magnesium absorption within subjects with and without chronic consumption of wheat dextrin.

ELIGIBILITY:
Inclusion Criteria:

- Subjects will be generally healthy Caucasian females aged 19 and older with no known abnormalities of gastrointestinal function, and taking no medications that might alter absorptive performance. BMI will be between 19 and 31 kg/m2

-

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Calcium Absorption | within 2-4 weeks
  The calcium load to be tested will be 300 mg calcium from calcium and vitamin D fortified TropicanaTM orange juice extrinsically labeled with ≈3-7 μCi of 45Ca. The labeled orange juice will be ingested as part of a light meal, served as breakfast, after an overnight fast.

SECONDARY OUTCOMES:
Magnesium absorption | within 2-4 weeks
  The magnesium load to be tested will be from calcium and vitamin D fortified TropicanaTM orange juice extrinsically labeled with 30 mg 26Mg. The labeled orange juice will be ingested as part of a light meal, served as breakfast, after an overnight fast.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Armas, MD, Principal Investigator — Creighton University